CLINICAL TRIAL: NCT00857220
Title: A Long Term, Open-Label, Safety Study of Eszopiclone in Children (6 to 11 Years) and Adolescents (12 to 17 Years) With Attention Deficit/Hyperactivity Disorder Associated Insomnia
Brief Title: Long Term Safety Study of Study Drug (Eszopiclone) in Children and Adolescents With ADHD -Associated Insomnia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 190-247
Record Dates: First submitted 2009-03-04; First posted 2009-03-06 (Estimated); Results first posted 2013-07-22 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-09

CONDITIONS: Insomnia; Attention Deficit Hyperactivity Disorder
Keywords: Hypnotic; Eszopiclone; Attention Deficit Hyperactivity Disorder; Insomnia; Children; Adolescent
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Attention Deficit Disorder with Hyperactivity | interventions — Eszopiclone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2mg eszopiclone (6-11yrs), 3mg eszopiclone (12-17yrs) (Experimental)
  Interventions: Drug: eszopiclone

INTERVENTIONS:
Drug: eszopiclone — One 2 mg tablet per day for 12 months
Drug: eszopiclone — one 3mg tablet per day for 12 months

SUMMARY:
A multicenter study to evaluate the safety of eszopiclone in children (6 11 years of age, inclusive) and adolescents (12 17 years of age, inclusive) with attention deficit/hyperactivity disorder (ADHD) associated insomnia.

DETAILED DESCRIPTION:
This is a multi center, open label, long term safety study in pediatric subjects 6 through 17 years of age, inclusive, with a diagnosis of ADHD associated insomnia. Subjects who complete Study 190 246 (Rollover subjects) and meet the study enrollment criteria will be allowed to participate in this long term safety study. Additionally, Treatment naïve subjects will be enrolled in this long term safety study in order to meet the overall subject enrollment objective of obtaining 100 subjects with 12 months of treatment. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Subject is male or female 6 17 years of age, inclusive, at the time of consent.
* Subject must have a diagnosis of ADHD as defined by DSM-IV criteria • The diagnosis for Rollover subjects will be taken from the Screening visit of Study 190 246. Treatment naïve subjects will have these assessments performed at the Screening visit.
* Subject must have documented ADHD associated insomnia, defined as the subject or subject's parent/legal guardian having reported repeated difficulty with sleep initiation (sleep latency >30 minutes) or consolidation (wake time after sleep onset > 45 minutes),>despite adequate age appropriate time and opportunity for sleep.
* Subject has either >30 minutes latency to persistent sleep (LPS) or >45 minutes wake time after sleep onset (WASO) demonstrated by PSG.
* Subject or subject's parent/legal guardian should have reported daytime functional impairment as a result of sleep problems.
* Subject or subject's parent/legal guardian should have reported attempted and failed behavioral interventions for sleep problems, including a regular bedtime and rise time.
* Subject's sleep disturbance must not be attributable to either the direct physiologic effect of a drug of abuse or misuse of a prescribed medication whether it is being used as intended or in an illicit manner.
* Female subjects ≥8 years of age must have a negative serum pregnancy test at screening
* Subject must be in good general health.
* Subject must be able to swallow tablets.
* If subjects are currently taking medication for ADHD, they must be on a stable dose and regimen for at least one month, and preferably for at least 3 months prior to the time of consent

Exclusion Criteria:

* Subject with weight <10th percentile for age and gender
* Subject has any clinically significant or unstable medical abnormality/illness
* Subject has a documented history of Bipolar I or II Disorder, major depression, conduct disorder, generalized anxiety disorder (other than obsessive-compulsive disorder) or any history of psychosis, as determined by medical or psychiatric history or as determined by clinical interview using the MINI-Kid at Visit 1.
* Subject has periodic limb movement >5 times per hour, as demonstrated on PSG.
* Subject has sleep disordered breathing, as demonstrated on PSG.
* Subject has another primary sleep disorder (or secondary sleep disorder that is causing clinical impairment or any other known or suspected medical or psychiatric condition that has affected or may affect sleep
* Subject has a history of circadian rhythm disorder or will travel across ≥3 time zones more than once during the study.
* Subject has organic brain disease, or a history of febrile seizures.
* Subject is, in the opinion of the investigator, at suicidal or homicidal risk.
* Female subject who is pregnant, lactating or planning to become pregnant.
* Subject is taking any psychotropic or disallowed medications,
* Subject has a history of severe allergies to more than 1 class of medications or multiple adverse drug reactions.
* Subject has a history of allergic reaction or has a known or suspected sensitivity to racemic zopiclone, eszopiclone, or any substance that is contained in the formulation.
* Subject has a history of alcohol or substance abuse within 3 months of study participation
* Subject has participated in any investigational study within 30 days prior to study entry or is currently participating in another clinical trial, except Study 190 246.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 304 (Actual)
Dates: Start 2009-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (89):
- United States (89):
  - REM Medical Clinical Research, Tucson, Arizona
  - Clinical Study Centers, LLC, Little Rock, Arkansas
  - AV Institute, Inc., Carson, California
  - Clinical Innovations, Inc., Costa Mesa, California
  - Behavioral Research Specialists, LLC, Glendale, California
  - Sun Valley Research Center, Imperial, California
  - Excell Research, Inc., Oceanside, California
  - North County Clinical Research (NCCR), Oceanside, California
  - Pacific Clinical Research Medical Group, Orange, California
  - SDS Clinical Trials, Inc., Orange, California
  - Clinical Innovations, Inc., Riverside, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Clinical Innovations, San Diego, California
  - Neuropsychiatric Research Center of Orange County, Santa Ana, California
  - Apex Research Institute, Santa Ana, California
  - Clinical Innovations, Inc., Santa Ana, California
  - Elite Clinical Trials, Inc., Wildomar, California
  - Delta Waves, Inc., Colorado Springs, Colorado
  - Sarkis Clinical Trials, Gainesville, Florida
  - MD Clinical, Hallandale, Florida
  - Amedica Research Institute, Inc., Hialeah, Florida
  - Behavioral Clinical Research Inc., Lauderhill, Florida
  - Behavioral Clinical Research, Inc., Lauderhill, Florida
  - Pediatric Neurology and Epilepsy Center, Loxahatchee Groves, Florida
  - Florida Clinical Research Center, LLC, Maitland, Florida
  - Scientific Clinical Research Inc., North Miami, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Florida Institute for Clinical Research, LLC, Orlando, Florida
  - DMI Research Inc., Pinellas Park, Florida
  - Florida Sleep Institute, Spring Hill, Florida
  - SomnoMedics, LLC, Tampa, Florida
  - Sleep Disorders Center of Georgia, Atlanta, Georgia
  - Northwest Behavioral Research Center, Roswell, Georgia
  - Mountain West Clinical Trials, Eagle, Idaho
  - Suburban Lung Associates, SC, Elk Grove Village, Illinois
  - Capstone Clinical Research, Libertyville, Illinois
  - AMR Baber Research, Inc., Naperville, Illinois
  - Sleep and Behavior Medicine Institute, Vernon Hills, Illinois
  - Davis Clinic, Indianapolis, Indiana
  - Goldpoint Clinical Research, LLC, Indianapolis, Indiana
  - Nassim, McMonigle, Mescia & Associates, New Albany, Indiana
  - Psychiatric Associates, Overland Park, Kansas
  - Brownsboro Park Pediatrics, Louisville, Kentucky
  - Pedia Research, LLC, Owensboro, Kentucky
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - Louisiana Research Associates, Inc., New Orleans, Louisiana
  - MD, Chevy Chase, Maryland
  - ActivMed Practices and Research, Haverhill, Massachusetts
  - Neurocare, Inc., Newton, Massachusetts
  - ActivMed Practices and Research, North Andover, Massachusetts
  - Neurobehavioral Medicine Group, Bloomfield Hills, Michigan
  - Clinical Nuerophysiology Services, PC, Sterling Heights, Michigan
  - Precise Research Centers, Flowood, Mississippi
  - Premier Psychicatric Research Institute, LLC, Lincoln, Nebraska
  - Midwest Children's Health Research Institute, Lincoln, Nebraska
  - Clinical Research Center of Nevada, Henderson, Nevada
  - Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada
  - Global Medical Institutes, LLC, Princeton, New Jersey
  - CRI Worldwide, LLC, Willingboro, New Jersey
  - NorthCoast Clinical Trials, Inc., Beachwood, Ohio
  - Neuro-Behavioral Clnical Research, Canton, Ohio
  - Cleveland Sleep Research Center, Middleburg Heights, Ohio
  - North Star Medical Research, LLC, Middleburg Heights, Ohio
  - Cutting Edge Research of Enid, Enid, Oklahoma
  - IPS Research Company, Oklahoma City, Oklahoma
  - Pahl Pharmaceutical Professionals, LLC, Oklahoma City, Oklahoma
  - SP Research, Oklahoma City, Oklahoma
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Eminence Research LLC, Oklahoma City, Oklahoma
  - Paradigm Research Professonals, LLP, Tulsa, Oklahoma
  - Tulsa Clinical Research, Tulsa, Oklahoma
  - Cyn3rgy Research, Gresham, Oregon
  - Oregon Center for Clinical Investigations, Inc., Portland, Oregon
  - Oregon Center for Clinical Investigations, Inc. (OCCI, Inc.), Salem, Oregon
  - CRI Worldwide, Philadelphia, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Holston Medical Group, Kingsport, Tennessee
  - Academy of Clinical Research, Arlington, Texas
  - Pillar Clinical Research, LLC, Dallas, Texas
  - InSite Clinical Research, DeSoto, Texas
  - Claghorn-Lesem Research Clinic, Ltd., Houston, Texas
  - Allegiant Clinical Research, Houston, Texas
  - MD, Houston, Texas
  - The Mech Center, Plano, Texas
  - Road Runner Research, San Antonio, Texas
  - Aspen Clinical Research, LLC, Orem, Utah
  - Alliance Research Group, Richmond, Virginia
  - Brighton Research Group, LLC, Virginia Beach, Virginia
  - Eastside Therapeutic Resource, Kirkland, Washington

REFERENCES:
- [Derived] Sangal RB, Blumer JL, Lankford DA, Grinnell TA, Huang H. Eszopiclone for insomnia associated with attention-deficit/hyperactivity disorder. Pediatrics. 2014 Oct;134(4):e1095-103. doi: 10.1542/peds.2013-4221. PMID 25266438

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The participant flow section includes all subjects randomized. The intent-to-treat (ITT) population consisted of all randomized subjects who had taken any study medication. One subject did not receive study medication.
Groups:
- 2mg Eszopiclone (6-11yrs), 3mg Eszopiclone (12-17yrs): Eszopiclone Overall
Period: Overall Study
Arm/Group | 2mg Eszopiclone (6-11yrs), 3mg Eszopiclone (12-17yrs)
Started | 304
Completed | 121
Not Completed | 183
Not completed — Adverse Event | 35
Not completed — Death | 1
Not completed — Lack of Efficacy | 11
Not completed — Lost to Follow-up | 30
Not completed — Physician Decision | 4
Not completed — Protocol Violation | 16
Not completed — Withdrawal by Subject | 67
Not completed — Clinical Hold | 6
Not completed — Site Closed | 5
Not completed — Miscellaneous | 8

BASELINE CHARACTERISTICS:
Arm/Group | 2mg Eszopiclone (6-11yrs), 3mg Eszopiclone (12-17yrs)
Number analyzed (Participants) | 303
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 303
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.2 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119
  Male | 184
Region of Enrollment [Number; unit: participants]
  United States | 303

OUTCOME MEASURES:

1. Primary Outcome: Overall Incidence of Adverse Events
Time Frame: 12 Months (from the 1st dose to the end of study)
Population: The intent-to-treat (ITT) population consisted of all enrolled subjects who had taken any study medication. One subject did not receive study medication
Measure: Number; unit: participants
Arm/Group | 2mg Eszopiclone (6-11yrs), 3mg Eszopiclone (12-17yrs)
Number analyzed (Participants) | 303
participants
  Subjects with at least 1 TEAE | 212
  Potentially-related TEAE | 138
  Severe TEAE | 10
  Serious TEAE | 4
  Fatal TEAE | 1
  Discontinued study due to TEAE | 34

2. Secondary Outcome: Overall Incidence of Skin Reactions: Number of Events
Time Frame: 12 Months (from the 1st dose to the end of study)
Population: Intent to treat population
Measure: Number; unit: Events
Arm/Group | 2mg Eszopiclone (6-11yrs), 3mg Eszopiclone (12-17yrs)
Number analyzed (Participants) | 303
Events | 17

3. Secondary Outcome: Overall Incidence of Skin Reactions: Number of Participant Affected
Time Frame: 12 Months (from the 1st dose to the end of study)
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | 2mg Eszopiclone (6-11yrs), 3mg Eszopiclone (12-17yrs)
Number analyzed (Participants) | 303
participants | 13

4. Secondary Outcome: Columbia-Suicide Severity Rating Scale (C-SSRS) Item Responses
Description: The C-SSRS is a physician-completed scale to assess any suicidal ideation and suicidal behavior. The C-SSRS contained questions about suicidal behavior and suicidal ideation. Subjects were placed into categories for suicidal behavior and for suicidal ideation based on their responses to various questions. Any suicidality was defined as suicidal behavior or suicidal ideation. The suicidal behavior categories were determined based on the response to the questions under suicidal behavior (Completed Suicide, Actual Attempt, Interrupted Attempt, Aborted Attempt, Preparatory Acts or Behavior).The suicidal ideation categories were determined by examining the response to 5 questions under suicidal ideation (Wish to be Dead, Nonspecific Active Suicidal Thoughts, Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act, Active Suicidal Ideation with Some Intent to Act, without Specific Plan, Active Suicidal Ideation with Specific Plan and Intent).
Time Frame: 12 Months
Population: Intent to treat population
Measure: Number; unit: Subjects
Arm/Group | 2mg Eszopiclone (6-11yrs), 3mg Eszopiclone (12-17yrs)
Number analyzed (Participants) | 303
Subjects
  Any Suicidality | 4 (1.3)
  Any Suicidal Behavior | 1 (0.3)
  Completed Suicide | 0 (0)
  Actual Attempt | 0 (0)
  Interrupted Attempt | 0 (0)
  Aborted Attempt | 1 (0.3)
  Preparatory Acts or Behavior | 0 (0)
  Any Suicidal Ideation | 4 (1.3)
  Wish to be Dead | 0 (0)
  Non-specific Active Suicidal Thoughts | 3 (1.0)
  Active Suicidal Ideation without Intent to Act | 0 (0)
  Active Suicidal Ideation w/ Some Intent to Act | 0 (0)
  Active Suicidal Ideation w/ Specific Plan | 1 (0.3)

5. Secondary Outcome: Change From Baseline in Coding Copy Subtest A or B, or Digit Symbol Substitution Test (DSST)at Month 12
Description: These tests are standardized information processing tasks to assess recognition and recoding of sensory information. The subject was given 90 seconds to complete as many substitutions of symbols as possible according to a code provided on top of the sheet. The Coding Copy Subtest A was used for subjects 6 to 7 years of age, the Coding Copy Subtest B was used for subjects 8 to 16 years of age, and the DSST was used for subjects 17 years of age. The DSST consists of rows containing small blank squares, each paired with a randomly assigned numbers 1-9. Above the rows is a key that pairs each number with a symbol. The subject must fill in the blank spaces with the matching symbol that is in the key. For the Subcopy tests the subject simply copies the symbol above each empty square. Scaled scores are used to account for age differences among test takers. Scaled scores range from 1 to 19, and higher scores indicate higher cognitive function.
Time Frame: Baseline and 12 Months (from the 1st dose to the end of study)
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: score
Arm/Group | 2mg Eszopiclone (6-11yrs), 3mg Eszopiclone (12-17yrs)
Number analyzed (Participants) | 303
score | 1.1 (6.1)

6. Secondary Outcome: Clinical Global Impression (CGI) Improvement Score as Assessed by Parent/Caregiver or Child at Month 12
Description: A 7-point scale was used for improvement with numeric values assigned to each of the responses: very much improved (1), much improved (2), minimally improved (3), no change (4), minimally worse (5), much worse (6), and very much worse (7).
Time Frame: Baseline and 12 Months (from the 1st dose to the end of study)
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 2mg Eszopiclone (6-11yrs), 3mg Eszopiclone (12-17yrs)
Number analyzed (Participants) | 303
units on a scale
  From Parent | 2.6 (1.4)
  From Child | 2.6 (1.5)

7. Secondary Outcome: Change From Baseline at Month 12 in Subjective Sleep Latency (SL)
Description: Sleep latency is the amount of time it takes to fall asleep after the lights have been turned off.
Time Frame: Baseline and 12 Months (from the 1st dose to the end of study)
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | 2mg Eszopiclone (6-11yrs), 3mg Eszopiclone (12-17yrs)
Number analyzed (Participants) | 303
Minutes | -18.1 (87.3)

8. Secondary Outcome: Change From Baseline in Child Behavior Checklist (CBCL)
Description: CBCL was completed by parents or guardians who saw the child in home-like settings. It includes several competence items, open-ended items for describing the child's illnesses, disabilities, concerns about the child, best things about the child, and several items to rate behavioral, emotional, and social problems. Responses are recorded on a Likert scale: 0 = Not True, 1 = Somewhat or Sometimes True, 2 = Very True or Often True. The checklist contains 120 questions. The standardized score is computed by determining the z-score by subtracting the mean for the subject's age group and gender from the raw score and then dividing this by the standard deviation for the subject's age group and gender. Next, multiply the zscore by 15 and then add 100. For activities scale, social scale, school scale, and total competence scale, higher values indicate higher competencies. For Internalizing problems, externalizing problems, and total problems, higher values indicate more problems.
Time Frame: Baseline and 12 Months (from the 1st dose to the end of study)
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 2mg Eszopiclone (6-11yrs), 3mg Eszopiclone (12-17yrs)
Number analyzed (Participants) | 303
units on a scale
  Activities scale standardized score | 1.04 (13.83)
  Social scale standardized score | 0.94 (14.29)
  School scale standardized score | 0.02 (11.49)
  Total competence standardized score | 1.02 (13.34)
  Internalizing problems standardized score | 0.19 (15.13)
  Externalizing problems standardized score | 0.29 (12.33)
  Total problems standardized score | 0.19 (14.16)

9. Secondary Outcome: Change From Baseline in Pediatric Daytime Sleepiness Scale (PDSS)at Month 12
Description: The PDSS total score ranges from a low of 0 where the individual is endorsing each item at the lowest level of daytime sleepiness to a high of 32 where the individual is endorsing each item at the highest level of daytime sleepiness.
Time Frame: Baseline and 12 Months (from the 1st dose to the end of study)
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 2mg Eszopiclone (6-11yrs), 3mg Eszopiclone (12-17yrs)
Number analyzed (Participants) | 303
units on a scale | -3.9 (6.0)

10. Secondary Outcome: Change From Baseline in Conners' Continuous Performance Test II (CCPT II)
Description: The CCPT-II is a computer-based 14-minute, visual-performance task. During an administration, respondents were required to press the space bar or click the mouse whenever any letter except the target letter appears on the screen. The speed at which the letters were presented varied during the administration. There were 6 blocks, with 3 sub-blocks, each containing 20 trials (letter presentations). The interstimulus intervals (ISIs) were 1, 2, and 4 seconds with a display time of 250 milliseconds. The order in which the different ISIs were presented varied between blocks. Conners' CCPT-II provides the following measures:% Omissions,% Commissions, Hit Reaction Time, Hit Reaction Time Standard Error,Variability of Standard Error, Detectability (d'), Response Style (beta), Perseverations, Hit Reaction Time Block Change (Vigilance Measure), Hit Standard Error Block Change (Vigilance Measure), Hit Reaction Time ISI change, and Hit Standard Error ISI Change, Confidence Index.
Time Frame: Baseline and 12 Months (from the 1st dose to the end of study)
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: percentage of score
Arm/Group | 2mg Eszopiclone (6-11yrs), 3mg Eszopiclone (12-17yrs)
Number analyzed (Participants) | 303
percentage of score
  Omissions % Percentile | 10.285 (29.390)
  Commissions % Percentile | -5.980 (29.332)
  Hit RT Percentile | 5.933 (27.606)
  Hit RT Std Error Percentile | 8.747 (30.776)
  Variability Percentile | 8.781 (32.543)
  Detectability (d') Percentile | -3.614 (33.471)
  Responsive Style (beta) Percentile | -3.614 (33.471)
  Perseverations % Percentile | 4.807 (25.389)
  Hit RT Block Change Percentile | 0.213 (33.614)
  Hit SE Block Change Percentile | -2.919 (36.037)
  Hit RT ISI Change Percentile | 8.070 (30.364)
  Hit SE ISI Change Percentile | 8.270 (35.780)
  Confidence Index | 8.471 (23.889)

11. Secondary Outcome: Change From Baseline at Month 12 in Subjective Wake Time After Sleep Onset (WASO)
Description: The sleep questionnaire, a Sponsor produced questionnaire used in previous eszopiclone studies, asked the subject or parent/guardian to report information about the subject's sleep and daytime functioning since the last visit. This questionnaire provided a subjective assessment of the subject's sleep over a predefined time period. WASO was assessed based on the responses to the sleep questionnaire.
Time Frame: Baseline and 12 Months (from the 1st dose to the end of study)
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | 2mg Eszopiclone (6-11yrs), 3mg Eszopiclone (12-17yrs)
Number analyzed (Participants) | 303
Minutes | -22.7 (70.5)

12. Secondary Outcome: Change From Baseline at Month 12 in Subjective Number of Awakening After Sleep Onset (NAASO)
Description: The sleep questionnaire, a Sponsor produced questionnaire used in previous eszopiclone studies, asked the subject or parent/guardian to report information about the subject's sleep and daytime functioning since the last visit. This questionnaire provided a subjective assessment of the subject's sleep over a predefined time period. NAASO was assessed based on the responses to the sleep questionnaire.
Time Frame: Baseline and 12 Months (from the 1st dose to the end of study)
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: Number of Awakenings
Arm/Group | 2mg Eszopiclone (6-11yrs), 3mg Eszopiclone (12-17yrs)
Number analyzed (Participants) | 303
Number of Awakenings | -0.8 (1.6)

13. Secondary Outcome: Change From Baseline at Month 12 in Subjective Total Sleep Time (TST).
Description: The sleep questionnaire, a Sponsor produced questionnaire used in previous eszopiclone studies, asked the subject or parent/guardian to report information about the subject's sleep and daytime functioning since the last visit. This questionnaire provided a subjective assessment of the subject's sleep over a predefined time period. TST was assessed based on the responses to the sleep questionnaire.
Time Frame: Baseline and 12 Months (from the 1st dose to the end of study)
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | 2mg Eszopiclone (6-11yrs), 3mg Eszopiclone (12-17yrs)
Number analyzed (Participants) | 303
Minutes | 45.3 (119.8)

14. Secondary Outcome: Change From Baseline in Pediatric Quality of Life Scale
Description: The SF-10™ Health Survey for Children is a 10-item care-giver completed assessment designed to measure children's health-related quality of life. The scale asked questions about the child's physical wellness, feelings, behavior, and activities at school and with family and friends. The SF-10 physical and psychosocial summary measures were scored such that higher scores indicated more favorable functioning. The Physical Summary Score is computed by summing values for questions 1, 2a, 2b, 3 and 5 and standardizing scores by normalizing to a total possible score of 0-100 with higher scores representing more positive indications. The Psychosocial Summary Score is computed by summing questions 4, 6, 7, 8, and 9 and standardizing scores by normalizing to a total possible score of 0-100 with higher scores representing more positive indications.
Time Frame: Baseline and 12 Months (from the 1st dose to the end of study)
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 2mg Eszopiclone (6-11yrs), 3mg Eszopiclone (12-17yrs)
Number analyzed (Participants) | 303
units on a scale
  Physical Summary Score | -1.31 (11.15)
  Psychosocial Summary Score | 2.14 (10.37)

ADVERSE EVENTS:
Time Frame: 12 Months
Description: The intent-to-treat (ITT) population consisted of all randomized subjects who had taken any study medication. The ITT population was used for all safety analyses.
Arm/Group | 2mg Eszopiclone (6-11yrs), 3mg Eszopiclone (12-17yrs)
Serious Adverse Events (participants affected / at risk) | 4/303
Other Adverse Events (participants affected / at risk) | 179/303
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2mg Eszopiclone (6-11yrs), 3mg Eszopiclone (12-17yrs) (N=303)
Drowning (General disorders) | 1 (1)
Viral Infection (Infections and infestations) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2mg Eszopiclone (6-11yrs), 3mg Eszopiclone (12-17yrs) (N=303)
Headache (Nervous system disorders) | 65 (123)
Dysgeusia (Nervous system disorders) | 42 (46)
Dizziness (Nervous system disorders) | 30 (35)
Somnolence (Nervous system disorders) | 15 (17)
Abdominal Pain Upper (Gastrointestinal disorders) | 19 (19)
Vomiting (Gastrointestinal disorders) | 15 (18)
Diarrhoea (Gastrointestinal disorders) | 13 (16)
Nausea (Gastrointestinal disorders) | 13 (14)
Toothache (Gastrointestinal disorders) | 9 (13)
Abdominal discomfort (Gastrointestinal disorders) | 7 (7)
Nasopharyngitis (Infections and infestations) | 20 (27)
Upper respiratory infection (Infections and infestations) | 12 (16)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 11 (14)
Influenza (Infections and infestations) | 10 (11)
Pharyngitis streptococcal (Infections and infestations) | 8 (8)
Urinary tract infection (Infections and infestations) | 6 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (18)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 (18)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 12 (14)
Pyrexia (General disorders) | 16 (20)
Influenza like illness (General disorders) | 6 (7)
Insomnia (Psychiatric disorders) | 10 (10)
Hallucination, visual (Psychiatric disorders) | 7 (8)
Contusion (Injury, poisoning and procedural complications) | 6 (6)

LIMITATIONS AND CAVEATS:
Designed to assess safety/tolerability. Efficacy endpoints evaluated w/ descriptive stats only, w/ no placebo group against which to assess the impact of therapy. ~40% completion rate typical for one year studies but limits interpretation of results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other